CLINICAL TRIAL: NCT05488626
Title: Daily Adaptive vs Non-Adaptive External Beam Radiation Therapy With Concurrent Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer: A Prospective Randomized Trial of an Individualized Approach for Toxicity Reduction (ARTIA-Lung)
Brief Title: Daily Adaptive Radiation Therapy: An Individualized Approach for Stage III Lung Cancer
Acronym: ARTIA-Lung
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Shifting patterns of care for the target population.
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-09
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stage III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adaptive Arm (Experimental): Subjects in this arm will receive their external beam radiotherapy on the Ethos Radiotherapy System version 2.0 with HyperSight cone beam computed tomography imaging, with daily online adaptation of their radiation dosimetry plan to account for day-to-day changes in the tumor and surrounding anatomical structures. All subjects will received standard concurrent chemotherapy and may receive adjuvant immunotherapy, if indicated.
  Interventions: Device: Adaptive Radiotherapy; Drug: Chemotherapy; Drug: Immunotherapy
- Non-Adaptive Arm (Active Comparator): Subjects in this arm will receive their radiotherapy using standard image-guided radiation therapy (IMRT) techniques. All subjects will receive standard concurrent chemotherapy and may receive adjuvant immunotherapy, if indicated.
  Interventions: Device: Non-Adaptive Radiotherapy; Drug: Chemotherapy; Drug: Immunotherapy

INTERVENTIONS:
Device: Adaptive Radiotherapy — Standard fractionation external beam radiotherapy (60-66 Gy in 2 Gy/fraction) with daily online adaptation.
  Arms: Adaptive Arm
Device: Non-Adaptive Radiotherapy — Standard fractionation external beam radiotherapy (60-66 Gy in 2 Gy/fraction) with daily image guidance.
  Arms: Non-Adaptive Arm
Drug: Chemotherapy — Concomitant chemotherapy per NCCN or other national guidelines.
Drug: Immunotherapy — Adjuvant immunotherapy per national or institutional guidelines.

SUMMARY:
This is a prospective multi-center randomized clinical trial designed to demonstrate that daily online adaptive radiotherapy with concomitant chemotherapy for stage III non-small cell lung cancer (NSCLC) will result in decreased acute respiratory and esophageal toxicity compared with non-adaptive radiotherapy with concomitant chemotherapy. The timepoint for this assessment will be 3 months following the end of radiotherapy and will use the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Histologically confirmed NSCLC
3. Clinical stage IIIA-IIIB (AJCC v8) disease who are either:

   1. Patients classified as non-operable by the treatment team
   2. Patients who refuse surgery
4. Clinical stage IIIC due to contralateral mediastinal lymph node involvement only (e.g., no contralateral hilar or any supraclavicular/cervical lymph node metastases). Mediastinal stations 2R and 4R are considered contralateral for patients whose primary tumor is within the left lung. Mediastinal stations 2L, 4L, 5, and 6 are considered contralateral for patients whose primary tumor is in the right lung.
5. Completed evaluation for metastatic disease with no distant metastases identified. Evaluation must include the following:

   1. History and physical examination within 30 days prior to enrollment.
   2. Whole body FDG PET-CT for staging within 60 days prior to enrollment
   3. Brain MRI or contrast enhanced CT within 60 days prior to enrollment.
6. ECOG performance status 0-2 and deemed clinically fit for chemoradiotherapy.
7. Age ≥18 years (or at least the local age of consent)
8. Patients must have normal organ and marrow function.
9. Serum creatinine ≤1.5 mg/dL within 60 days prior to enrollment.
10. Measurable disease must be present.
11. Negative urine or serum pregnancy test within 14 days prior to enrollment for women of childbearing potential.

Exclusion Criteria:

1. Contralateral hilar or any supraclavicular/cervical lymph nodes.
2. Baseline grade ≥3 dyspnea, or cough, or dysphagia.
3. Prior invasive non-skin malignancy unless disease free for a minimum of 3 years.
4. History of prior RT to the thorax.
5. Severe imaging artifact that, in the view of the local investigator, would preclude accurate identification of the thoracic anatomy and tumor targets on the cone beam CT (e.g., artifact created implanted cardiac device in proximity to the targets).
6. Evidence of malignant pleural effusion, defined as either FDG PET avidity within effusion fluid or presence of malignant cells identified by cytology of thoracentesis fluid.
7. Severe active chronic obstructive pulmonary disease or respiratory illness other than NSCLC precluding study therapy.
8. Hospitalization for chronic obstructive pulmonary disease or respiratory illness other than NSCLC within 1 year prior to study enrollment.
9. Women of childbearing potential and sexually active women not willing or able to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | From randomization to 90 days after completion of chemoradiotherapy
  Composite rate of any increase in cough, or dyspnea, or dysphagia scores by 1+ using PRO-CTCAE.

SECONDARY OUTCOMES:
Lung cancer specific quality of life | From randomization to 12 months after completion of chemoradiotherapy
  Results from the FACT-L questionnaire
Global quality of life | From randomization to 12 months after completion of chemoradiotherapy
  Results from the EQ-5D-5L questionnaire
Normal lung tissue radiation exposure | End of external beam radiation treatment (approximately 2 months from randomization)
  The percentage of normal lung tissue volume that receives radiation of 20 Gy or more over the course of radiation treatment.
Mean normal tissue doses | End of external beam radiation treatment (approximately 2 months from randomization)
  Mean dose delivered to the heart, esophagus and normal lung tissue over the course of radiation treatment.
Overall response rate | 3 months, 6 months and 12 months after completion of chemoradiotherapy
  Frequency of complete and partial tumor response as determined on chest imaging using RECIST v1.1
Local progression | 12 months after completion of chemoradiotherapy
  Physician report of progression determined by imaging or clinical evaluation
Radiation pneumonitis | 12 months after completion of chemoradiotherapy
  CTCAE v.5.0 grade 2+ pneumonitis
Healthcare resource utilization | From the start of radiation treatment to 12 months after completion of chemoradiotherapy.
  Hospitalizations, emergency department visits, advanced medical or imaging procedures associated with the treatment of CTCAE grade 2+ adverse events related to EBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McDonald, MD, Principal Investigator — University of Alabama at Birmingham; Dennis Stanley, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No